CLINICAL TRIAL: NCT07280442
Title: Effectiveness of a Sodium Hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash for the Treatment of Symptomatic Oral Lichen Planus. A Randomized Clinical Trial
Brief Title: Effectiveness of a Sodium Hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash for the Treatment of Symptomatic Oral Lichen Planus
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 25/288-E
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus; RCT; OPMD; treatment; topical treatment; Sh-Oligopeptide-85 SP Mouthwash; Sodium hyaluronate 0.01%
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash (Experimental): Patients in the study group will be instructed to use 20 mL of Tectum-11® mouthwash after toothbrushing three times a day for 2 minutes. This procedure will be repeated daily throughout the 4-week treatment period. Patients will be asked not to eat or drink for 30 minutes after using the mouthwash.
  Interventions: Combination Product: Sodium hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash
- placebo mouthwash (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: Sodium hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash — Patients in the study group will be instructed to use 20 mL of Tectum-11® mouthwash after toothbrushing three times a day for 2 minutes. This procedure will be repeated daily throughout the 4-week treatment period. Patients will be asked not to eat or drink for 30 minutes after using the mouthwash.
  Arms: Sodium hyaluronate 0.01% and Sh-Oligopeptide-85 SP Mouthwash
Other: Placebo — Patients in the placebo group will use 20 mL of the placebo mouthwash after toothbrushing three times a day for 2 minutes. This procedure will be repeated daily throughout the 4-week treatment period. Patients will be asked not to eat or drink for 30 minutes after using the mouthwash.
  Arms: placebo mouthwash

SUMMARY:
Annex 1. Patient Information and Informed Consent for the Study Study Title: Effectiveness of a sodium hyaluronate 0.01% and Sh-Oligopeptide-85 SP mouthwash for the treatment of symptomatic oral lichen planus: a randomized clinical trial.

Principal Investigator: Dr. Rosa Mª López-Pintor Muñoz, Associate Professor, Department of Clinical Dental Specialties, Faculty of Dentistry, Complutense University of Madrid.

Dear Sir/Madam, Participants are invited to take part in a study evaluating the effectiveness of a mouthwash designed to reduce oral lichen planus-related lesions and pain.

Study Objective The primary aim of this study is to evaluate and compare the effect of Tectum mouthwash (containing sodium hyaluronate and Sh-Oligopeptide-85) versus a corticosteroid mouthwash (provided at no cost to participants) in reducing pain and lesion size.

Eligible participants with oral lichen planus and associated discomfort will receive either Tectum mouthwash or a corticosteroid mouthwash to use after toothbrushing for the first two weeks three times daily, twice daily in the third week, and once daily in the fourth week of treatment.

Participants will be randomly assigned to receive either Tectum mouthwash or the corticosteroid mouthwash through a process comparable to a coin toss. Treatment allocation will be blinded. Neither participants nor the attending clinician will know which treatment is being administered. Participants must use the assigned mouthwash for 4 weeks according to the clinician's instructions and attend visits at the Faculty of Dentistry at 1, 2, 3, and 4 weeks to assess improvement.

At the first visit, a series of data will be recorded, and oral lichen planus lesions and pain will be assessed. The same variables will be evaluated at 1, 2, 3, and 4 weeks to determine treatment effectiveness. Participants will also complete two questionnaires assessing pain intensity and the impact of symptoms on quality of life. During the 4-week treatment period, the use of any other mouthwashes will not be permitted, and antibiotics or anti-inflammatory medications may not be used.

The investigational mouthwash is already marketed and has been used to treat conditions such as oral mucositis and xerostomia with favorable results; therefore, potential benefit in oral lichen planus is anticipated.

If pain occurs, 400 mg ibuprofen may be taken every 8 hours as needed. If ibuprofen is taken, each dose should be recorded and reported to the attending healthcare professional.

Voluntary Participation Participation is entirely voluntary, and non-participation is permitted. Participants may withdraw at any time without providing an explanation and without any disadvantage to clinical care. Refusal to participate or withdrawal will not affect the relationship between participants and the institution.

Study Procedures The dentist providing care in the Diploma of Specialization in Oral Medicine will invite eligible individuals to participate and will provide detailed instructions. The attending dentist will request completion of a questionnaire containing study-required information. If participation is accepted, lesions will be assessed, and questionnaires will be completed.

The attending dentist will instruct participants on product use: three times daily during weeks 1 and 2, twice daily during week 3, and once daily during week 4. Follow-up appointments at 1, 2, 3, and 4 weeks will be scheduled to evaluate the same variables and to repeat the questionnaires.

Risks This study does not present additional risks beyond routine care. Improvement may not occur with use of the mouthwash. Response to corticosteroids and to the investigational treatment may vary.

Confidentiality Confidentiality will be maintained. All information collected during this research will be treated as privileged and documented in coded format. Participants have the right to access and rectify personal data at any time, as established by Organic Law 3/2018 of December 5 on the Protection of Personal Data and Guarantee of Digital Rights. In accordance with data protection regulations, consent may be revoked and rights of access, modification, opposition, and deletion of data may be exercised. Rights to limit the processing of inaccurate data, request a copy of the data, or request transfer of data to a third party (portability), as applicable, may also be exercised.

To exercise these rights, contact may be made with the principal investigator (Dr. Rosa Mª López-Pintor Muñoz, Department of Clinical Dental Specialties, Faculty of Dentistry, Complutense University of Madrid). Participants may also contact the Spanish Data Protection Agency if concerns are not resolved satisfactorily.

Participant identity and any information that could identify a participant will not be disclosed.

ELIGIBILITY:
Patients must meet the following inclusion criteria:

1. Patients aged ≥18 years.
2. Patients with a clinical and histological diagnosis of OLP according to the criteria of the American Academy of Oral and Maxillofacial Pathology (Cheng et al., 2016).
3. Symptomatic patients, i.e., those presenting atrophic-erosive or ulcerative OLP lesions.
4. Patients with a VAS score ≤ 6.

Exclusion criteria will be:

1. Pregnant or breastfeeding women.
2. Allergy to the components of the Tectum-11® mouthwash.
3. Patients receiving corticosteroids, immunosuppressants, hydroxychloroquine, or retinoids at the time of recruitment.
4. Patients with lichenoid lesions: drug-induced lichenoid reactions, contact lichenoid lesions, or graft-versus-host disease.
5. Use of topical corticosteroids within the previous 4 weeks or systemic treatment within the previous 8 weeks.
6. Use of other mouthrinses for plaque control.
7. Patients unwilling to sign the informed consent form.
8. Patients with a VAS score > 6.

The presence of any of the following criteria will lead to withdrawal of the participant from the study:

1. Failure to attend follow-up visits.
2. Occurrence of adverse events deemed clinically relevant by the investigator.
3. The patient reports that they no longer wish to participate in the study.
4. Development of oral or systemic lesions that meet any of the exclusion criteria.
5. Non-adherence to the treatment regimen, defined as failure to follow the protocol for more than two consecutive weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-12-17 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | at baseline, 7days, 14days, 21 days, 28days
  pain form 0 to 10 (0: no pain; 10: worst pain imaginable)

SECONDARY OUTCOMES:
Reticular Erosive Ulcerative score (REU), (from 0 to 115). The higher the score, the greater the severity | baseline, 7days, 14days, 21days, 28days
  To assess the appearance and severity of the lesions, the REU scoring system, validated for OLP, will be used. This grading system assigns a site-specific score according to the type of lesion present (reticular, erosive, or ulcerative), which are weighted in a final formula to determine a single overall lesion score for each patient. The anatomical sites are: upper and lower labial mucosa, right buccal mucosa, left buccal mucosa, soft palate, hard palate, floor of the mouth, dorsal tongue, ventral tongue, maxillary gingiva, and mandibular gingiva. The site-specific scoring will be as follows:
  Reticular or hyperkeratotic lesions:
  0: No white lesions
  1: Presence of striated lesions or hyperkeratotic papules
  Erythematous or erosive lesions:
  0: No lesion
  1. Lesion <1 cm²
  2. Lesion 1-3 cm²
  3. Lesion >3 cm²
  Ulcerative lesions:
  0: No lesion
  1. Lesion <1 cm²
  2. Lesion 1-3 cm²
  3. Lesion >3 cm² The total score across the 10 sites will be calculated using the followi
Oral Health Impact Profile 14 (OHIP-14) From 0 to 56. The higher the OHIP-14 score, the worse the oral health-related quality of life | baseline, 76days, 14days,21days,28days
  To assess the impact of OLP on the patient's oral health-related quality of life, the Oral Health Impact Profile (OHIP-14) will be used. This instrument evaluates seven dimensions:
  Functional limitation Physical pain Psychological discomfort Physical disability Psychological disability Social disability Handicap
  The OHIP-14 comprises 14 items, each scored on a 5-point Likert scale:
  0 = Never
  1. = Hardly ever
  2. = Occasionally
  3. = Fairly often
  4. = Very often

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Especialidades Clínicas Odonotlógicas, Facultad de Odontología, Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided